CLINICAL TRIAL: NCT02979821
Title: A Phase II Study to Assess Efficacy of Pan-HER Inhibitor (HM781-36B, Poziotinib) in Stage IV Lung Adenocarcinoma With HER2 Mutation
Brief Title: Poziotinib in Stage IV Lung Adenocarcinoma With HER2 Mutation (KASTT001)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Korean Association for the Study of Targeted Therapy (Other)
Collaborators: Konkuk University Medical Center (Other); Kyungpook National University Hospital (Other); Kosin University Gospel Hospital (Other); Chonnam National University Hospital (Other); Chungnam National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PZT1401
Record Dates: First submitted 2016-11-24; First posted 2016-12-02 (Estimated); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: HER2 Gene Mutation; Adenocarcinoma Lung Stage IV
Keywords: pan-HER inhibitor
MeSH Terms: conditions — Adenocarcinoma of Lung | interventions — HM781-36B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Poziotinib (Experimental): The study drug(poziotinib) will be administered orally as one 12 mg tablet once a day until disease progression or manifestation of unacceptable toxicity. The initial dose of the study drug 12 mg daily can be reduced to 8 mg once daily according to dose reduction criteria.
  Interventions: Drug: Poziotinib

INTERVENTIONS:
Drug: Poziotinib — A cycle of study treatment is defined as 28 days.
  Other Names: NOV120101

SUMMARY:
In this trial, treatment efficacy and safety of Poziotinib will be assessed in patients with stage IV lung adenocarcinoma harboring HER2 mutation.

DETAILED DESCRIPTION:
This study is designed to be multi-center, open-label, single-arm, prospective, phase II trial of patient with stage IV lung adenocarcinoma with HER2 mutation who have not received prior EGFR-TKI. Approximately 47 patients will be enrolled into the trial, and expected study duration is 36 months from IRB and Korea: MFDS approval date.

The study drug(poziotinib) will be administered orally as one 12 mg tablet once a day until disease progression or manifestation of unacceptable toxicity. The initial dose of the study drug 12 mg daily can be reduced to 8 mg once daily according to dose reduction criteria in protocol. A cycle of study treatment is defined as 28 days.

ELIGIBILITY:
Inclusion Criteria:

1. lung adenocarcinoma, stage IV
2. Patients with HER2 mutation by sequencing

   - Confirmed triple-negative patients with remnant tumor DNA
3. Patients who have histories of previous exposure to at least one more systemic chemotherapies (not EGFR-TKI)
4. ECOG performance status 0~2
5. Patient with at least one measurable lesions according to RECIST
6. Patients who have proper organ functions as follows

   * Neutrophil count: > 1,500/uL
   * Platelet count: > 100,000/uL
   * Hb: > 9.0g/dL
   * AST/ALT : < 2.0 x upper normal limit
   * Bilirubin: < 1.25 x upper normal limit
   * Serum creatinine : < upper normal limit

Exclusion Criteria:

1. Expected lie expectancy < 3 months
2. CNS metastasis or spinal cord compression which were not treated with operation and/or radiation therapy(but, Patient with medically stable condition after operation and/or radiation therapy, or without symptomatic metastasis of brain in accordance with the investigator's judgment could participate in the study)
3. Patients who have severe or unstable systemic disease in accordance with the investigator's judgment(ex, unstable or uncompensated respiratory, cardiac, hepatic or renal disease)
4. Patients who have histories of previous exposure to EGFR-TKI

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate; ORR including rage of CR&PR | through study completion (3 years)
  It will be assessed on based of RECIST 1.1.

SECONDARY OUTCOMES:
Time to progression, TTP | through study completion (3 years)
  from first IP administration to date of first documented progression

CONTACTS AND LOCATIONS:
Overall Officials: Kye-Young, Lee, MD, PhD, Principal Investigator — Kunkok University Medical Center
Locations (1):
- Korean Association for the Study of Targeted Therapy, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided